CLINICAL TRIAL: NCT05660486
Title: The Effects of Aromatherapy on Anxiety Prior to Ultrasound Guided Musculoskeletal Procedures: A Randomized Controlled Trial
Brief Title: Aromatherapy Effect on Anxiety Prior to Ultrasound Guided Musculoskeletal Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Tricia Prince, Assistant Professor of clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20220850
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy group (Experimental): Participants in this group will receive, lavender essential oil applied to their surgical mask for 5 minutes prior to scheduled standard of care ultrasound guided musculoskeletal procedure.
  Interventions: Other: Aromatherapy
- Placebo group (Placebo Comparator): Participants in this group will receive water applied to their surgical mask for 5 minutes prior to scheduled standard of care ultrasound guided musculoskeletal procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — Participants in this group will receive 2-3 drops of 100% pure Lavandula angustifolia essential oil applied to a surgical mask pre-procedure for aromatherapy.
  Arms: Aromatherapy group
Other: Placebo — Participants in this group will receive 2-3 drops of water applied to a surgical mask pre-procedure.
  Arms: Placebo group

SUMMARY:
The goal of this study is to evaluate the effect of lavender essential oil on pre-procedure anxiety for patients undergoing ultrasound guided musculoskeletal procedures

ELIGIBILITY:
Inclusion criteria: Adults ages 18-85. Those undergoing ultrasound guided musculoskeletal procedures including joint, tendon, bursa, or periarticular structure injection/ aspiration. Proficient with English.

Exclusion criteria:

Patients currently on benzodiazepine anxiolytic therapy Those with significantly impaired sense of smell Allergy/aversion to lavender essential oils Patients with asthma Patients with history of migraines Patients with any other condition that, in the opinion of the investigator, would compromise the well-being of the patient or prevent the patient from meeting or performing study requirements Adults unable to consent Individuals who are not yet adults Pregnant women Prisoners

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Anxiety state as measured by VASA | Up to 10 minutes after aromatherapy administration
  The Visual Analogue Scale for Anxiety (VASA) has scales ranging from 0 indicating "no anxiety" to 10 indicating "high anxiety"

SECONDARY OUTCOMES:
Number of participants with an aborted ultrasound guided procedure | Up to 60 minutes post aromatherapy administration
  Number of participants with an aborted ultrasound guided procedure due to intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Prince, DO, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No